# Insights from Spinal Cord Injury Clinical Trials Patients: A Review of Clinical Trial Experiences

Informed Consent Form (ICF) For <u>Power Clinical Trial's</u> Spinal Cord Injury Clinical Trial

Date: April 13, 2023

Examining the Informed Consent Form's Function in Clinical Trials

Clinical studies must include an informed consent form to ensure that potential participants are fully informed of the study's procedures, risks, and benefits before deciding to participate. The form is divided into two sections: a Patient Information Sheet outlining the study's main components and a Certificate of Consent attesting to the participant's free consent to participate. Although signing the form does not signify a participant's waiver of rights or commitment to further participation, it is crucial to preserve a copy for your records.

Understanding the Importance of Spinal Cord Injury Clinical Trials

Spinal cord injury (SCI) is a condition that occurs when the spinal cord is damaged, either partially or completely, resulting in a loss of sensory, motor, or autonomic function below the level of injury. The injury can be caused by trauma, such as a car accident or a fall, or by diseases such as cancer or infections.

SCI can have a devastating impact on a person's life, leading to paralysis, loss of bladder and bowel control, difficulty breathing, and chronic pain. There is currently no cure for SCI, and treatment options are limited to managing symptoms and preventing further damage.

Clinical trials for SCI are important because they offer a potential avenue for developing new treatments and improving outcomes for people with SCI.

To ensure that clinical trial participation rates adequately represent the broader community of patients with spinal cord injury, it is crucial to understand and address the factors that may contribute to underrepresented groups having lower participation rates. This clinical study aims to identify and understand these factors and develop effective strategies for increasing participation rates in future clinical trials.

We believe that by identifying and understanding the reasons for low participation rates in underrepresented groups, we can develop better plans to increase participation rates in upcoming clinical trials. It is important to note that participation in this clinical trial is entirely voluntary, and participants are free to withdraw at any time without penalty. Participants face minimal risk during the study's primary procedures, which involve completing surveys and follow-up calls. We encourage prospective participants to carefully review the consent form and consult with their loved ones, trusted advisers, and medical professionals before making a decision.

## Clinical Trial Methodology

The primary objective of this clinical trial is to gather valuable insights into the disease and help develop better treatments in the future. As an observational study, your current treatment plan will remain unchanged, and no intervention will be performed. If you choose to participate, the researcher will conduct interviews to collect data and improve their understanding of the disease's impact on patients' lives. It is important to note that the researcher cannot diagnose or recommend any treatment. Participation in this study is entirely voluntary, and you are free to withdraw at any time without any consequences. By taking part in this clinical trial, you will be contributing to the advancement of knowledge in this field, which could potentially benefit other patients in the future.

Understanding Patient Motivations in Clinical Trials for Spinal Cord Injury

Our research project focuses on patients who are currently participating in a clinical trial for spinal cord injury. We aim to gain insights into the motivations behind patients' decisions to take part in such studies and the factors that influence their decision to continue or withdraw from the trial.

Participation in this study is entirely voluntary, and it will not impact your current treatment plan. We will conduct interviews to collect data, which will be used to develop better strategies to improve patient recruitment and retention in future clinical trials.

Your input is crucial in helping us understand the perspectives and experiences of patients who participate in clinical trials for spinal cord injury. If you decide to take part, you can withdraw from the study at any time without any negative consequences.

#### **Exploring Options for Spinal Cord Injury Clinical Trials**

Access to numerous interventional clinical studies is available to patients with spinal cord injuries. This study sets itself apart by being strictly observational in nature and without requiring involvement in any specific treatment strategy.

It is crucial to highlight that there are other additional research possibilities available. Although we are unable to list them all, interested parties should visit clinicaltrials.gov for a full list of <u>spinal cord injury</u> studies or Power's website to learn more about their alternatives and active <u>spinal cord injury clinical trials</u> near you.

### **Explore Studies on Diversity in Clinical Trials**

If you are looking to learn more about diversity and representation in clinical trials, we suggest delving into published studies on the topic.

<u>Unger, Joseph M., Dawn L. Hershman, Mark E. Fleury, and Riha Vaidya. "Association of patient comorbid conditions with cancer clinical trial participation." *JAMA oncology* 5, no. 3 (2019): 326-333.</u>

Chen Jr, Moon S., Primo N. Lara, Julie HT Dang, Debora A. Paterniti, and Karen Kelly. "Twenty years post-NIH Revitalization Act: Enhancing minority participation in clinical trials (EMPaCT): Laying the groundwork for improving minority clinical trial accrual: Renewing the case for enhancing minority participation in cancer clinical trials." *Cancer* 120 (2014): 1091-1096.

#### Patient Statement

I confirm that I have been chosen to participate in a clinical trial for patients with spinal cord injuries. I have carefully read and understood the consent form, and any queries or concerns I had have been addressed to my satisfaction. I willingly agree to take part in

| secure. | | |
|---|---|---|
| Patient's Signature | | |
| Name of Patient | Signature of Patient | <br>Date |
| Declaration of Person | Getting Consent | |
| study, I ensured that the p<br>involved explaining the co<br>allowing sufficient time for<br>agreed to participate in the | for obtaining the participant's con<br>articipant fully understood all aspe<br>ntents of the consent form in a cle<br>any questions to be asked. I conf<br>e study voluntarily, without any coo<br>y. Lastly, I provided the participant | ects of the research. This ear and concise manner and firm that the participant ercion or undue influence |
| Signature of the Perso | n Getting Consent | |
| Name | Signature | <br>Date |

this study, and I am aware that my participation is voluntary, and I can withdraw from the study at any time without consequences. Furthermore, I understand that my personal data will be kept confidential, and any data collected during the research will be kept